CLINICAL TRIAL: NCT02874339
Title: High Flow Nasal Oxygen Versus VNI for Emergency Department Treatment of Acute Hypercapnic Cardiogenic Pulmonary Edema With Respiratory Failure: a Multicenter Randomized Non Inferiority Trial
Brief Title: High Flow Nasal Oxygen Versus VNI in Acute Hypercapnic Cardiogenic Pulmonary Edema
Acronym: OPTICAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9675; 2016-A00349-42 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2016-07-28; First posted 2016-08-22 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Acute Cardiogenic Pulmonary Edema; Hypercapnic Respiratory Failure
Keywords: Acute cardiogenic pulmonary; Respiratory failure; Hypercapnia; High flow nasal oxygen; Non invasive ventilation; Emergency department
MeSH Terms: conditions — Respiratory Insufficiency; Hypercapnia; Emergencies | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optiflow Group (Experimental): High flow nasal oxygen therapy
  Interventions: Device: High flow nasal oxygen therapy
- NIV group (Active Comparator)
  Interventions: Device: Non invasive ventilation

INTERVENTIONS:
Device: High flow nasal oxygen therapy — In the optiflow group, oxygen will be administered through a heated humidifier (Airvo 2, Fisher and Paykel healthcare) and applied through large bore binasal prongs. Initial gas flow rate will be set at of 60 l/min and adjusted to 40-50 l/min based on patient's tolerance. FiO2 will be adjusted to maintain an SpO2 ≥ 92%. Initial temperature will be set at 37° and reduced according to patient's tolerance.
  Other Names: Optiflow TM
  Arms: Optiflow Group
Device: Non invasive ventilation — In the NIV group, NIV will be delivered through a face mask connected to a ventilator with pressure support applied in a noninvasive ventilation mode. The Pressure-support level will be adjusted to obtain an expired tidal volume of 6-8 ml/kg of predicted body weight and a respiratory rate of 25-30 b/min. PEEP (range 5-10 cm of water) and FiO2 will be adjusted to maintain an SpO2 ≥92% and to patient's comfort.
  Arms: NIV group

SUMMARY:
The purpose of this study is to determine whether high flow nasal oxygen (HFNO) therapy is non inferior to non invasive ventilation (NIV) in the immediate treatment of patients with acute hypercapnic cardiogenic pulmonary edema associated with respiratory failure in the emergency department.

DETAILED DESCRIPTION:
Prospective multicenter study including ED patients with a suspected diagnosis of acute hypercapnic pulmonary edema with respiratory failure who require NIV according to the joint recommendations from the French society of anaesthesia and intensive care and the French society for intensive care.

Patients will be randomly assigned to NIV or high flow nasal oxygen therapy, with stratification on center and severity of hypercania.

Assigned Treatment will be administered during at least one session of 1hr and resumed as needed based on the patient's signs of respiratory distress and blood gas results Repeat evaluation of arterial blood gases, clinical parameters and dyspnea will be performed before and after the first and second hour of treatment according to current recommendation from the French society of anesthesia and intensive care medicine (SFAR).

ELIGIBILITY:
Inclusion criteria:

* Asuspected diagnosis of acute pulmonary edema presenting with any of the following criteria:
* Dyspnea (orthopnea or a worsening of dyspnea according to NYHA criteria)-Respiratory rate >20 b/min
* Bilateral crepitant rales at pulmonary auscultation
* Pulmonary infiltrate on chest X-ray
* Signs of respiratory failure or any of the following clinical, laboratory or or radiology signs:

  * Use of accessory respiratory muscles
  * Paradoxical abdominal movement
  * Cardiomegaly (cardiothoracic ratio >0.5)
  * Hypertensive crisis
  * PaO2/FiO2 <= 300 mmHg breathing O2> 8L/min or PaO2 <= 63mmHg breathing room air.
* Hypercapnia (PaCO2>45)

Exclusion criteria:

* Chronic respiratory disease or associated dyspnea from non cardiac origin,
* Fever (>38,5°), sepsis or ongoing infection,
* Contra-indication to NIV,
* Treatment with NIV or CPAP prior to inclusion, including prehospital treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-10-26; Primary Completion 2018-10 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a normalized PaCO2 | 1hr of treatment
  (PaCO2 equal or lower than 45 mmHg)

SECONDARY OUTCOMES:
Blood gas parameters | 1hr
  Blood gas parameters will be measured from standard laboratory arterial blood gas analysis
Blood gas parameters | 2hr
  Blood gas parameters will be measured from standard laboratory arterial blood gas analysis
Blood gas parameters | End of management (before discharge from ER)
  Blood gas parameters will be measured from standard laboratory arterial blood gas analysis
Patient's dypnea | 1hr
  Dyspnea will be assessed by the emergency physician based on patient's use of accessory respiratory muscles, and measured using a 5-point likert scale.
  Dyspnea score will be recorded by the patient using a Modified Borg scale for dyspnea
Patient's dypnea | 2hr
  Dyspnea will be assessed by the emergency physician based on patient's use of accessory respiratory muscles, and measured using a 5-point likert scale.
  Dyspnea score will be recorded by the patient using a Modified Borg scale for dyspnea
Patient's dypnea | End of management (before discharge from ER)
  Dyspnea will be assessed by the emergency physician based on patient's use of accessory respiratory muscles, and measured using a 5-point likert scale.
  Dyspnea score will be recorded by the patient using a Modified Borg scale for dyspnea
Patient's comfort | 1hr
  Comfort score will be recorded by the patient using a visual analog scale from 0 to 10 for comfort
Patient's comfort | 2hr
  Comfort score will be recorded by the patient using a visual analog scale from 0 to 10 for comfort
Patient's comfort | End of management (before discharge from ER)
  Comfort score will be recorded by the patient using a visual analog scale from 0 to 10 for comfort
Endotracheal intubation | 7 day and 1 month follow up
Mortality | 7 day and 1 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha Sebbane, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided